CLINICAL TRIAL: NCT02134873
Title: Sucrose Practices for Pain in Neonates: A Program of Research: Part A (Trial 1 and 2): Determining the Minimally Effective Dose of Sucrose for Procedural Pain in Infants
Brief Title: Sucrose Practices for Pain in Neonates
Acronym: SPiN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Bonnie Stevens, Dr. Bonnie Stevens, RN, PhD, Signy Hildur Eaton Chair in Paediatric Nursing Research, Associate Chief of Nursing Research, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1000038052
Record Dates: First submitted 2014-05-05; First posted 2014-05-09 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Pain
Keywords: Pain; Pain management; Hospitalized; Infants; Sucrose
MeSH Terms: conditions — Pain; Agnosia | interventions — Sucrose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- 0.1ml 24% sucrose concurrent opioids (Active Comparator): 0.1ml 24% sucrose concurrent opioids
  Interventions: Other: sucrose
- 0.5ml 24% sucrose concurrent opioids (Active Comparator): 0.5ml 24% sucrose concurrent opioids
  Interventions: Other: sucrose
- 1.0ml 24% sucrose concurrent opioids (Active Comparator): 1.0ml 24% sucrose concurrent opioids
  Interventions: Other: sucrose
- 0.1ml 24% sucrose no opioids (Active Comparator): 0.1ml 24% sucrose no opioids
  Interventions: Other: sucrose
- 0.5ml 24% sucrose no opioids (Active Comparator): 0.5ml 24% sucrose no opioids
  Interventions: Other: sucrose
- 1.0ml 24% sucrose no opioids (Active Comparator): 1.0ml 24% sucrose no opioids
  Interventions: Other: sucrose

INTERVENTIONS:
Other: sucrose — Sucrose will be administered by a research nurse experienced in neonatal intensive care using a standardized procedure and timing consistent with policies in the participating units, including: (a) administering sucrose 2 minutes prior to the heel lance to ensure peak effects; (b) giving the total volume of sucrose drop by drop via syringe on the anterior surface of the tongue, as tolerated, over a period of up to 1 minute to allow for individual infant swallowing rates and to ensure analgesic effects are sustained during the heel lance procedure; and (c) offering a pacifier for non-nutritive sucking (NNS) immediately following sucrose administration.
  Other Names: Brand name = Tootsweet

SUMMARY:
Recent studies show that babies in hospital undergo an average of 4 to 5 painful procedures, such as heel lances, every day. Sucrose (sugar water) has been shown to be effective for reducing pain during invasive procedures and is a standard of care for painful procedures. The purpose of this study is to see what is the least amount of sucrose that can be given to a baby to reduce pain during procedures.

DETAILED DESCRIPTION:
Infants in the NICU receive an average of 4 - 5 painful procedures daily for diagnostic and therapeutic purposes; less than half receive interventions to manage pain. Both immediate and long term effects of unmanaged pain in these vulnerable infants have been reported, including impaired brain development. To ensure optimal outcomes for hospitalized infants in NICUs, there is a crucial need to minimize procedural pain and its associated consequences. Multiple clinical trials have identified sucrose as an effective strategy for reducing procedural pain in infants. Despite its inclusion in neonatal pain guidelines, standards, and consensus statements sucrose has been inconsistently used. The under-utilization of sucrose may be explained by knowledge gaps in relation to the minimally effective dose and the influence of concurrent opioid analgesia, as well as the short and long-term effects of repeated administration. Once infants in the NICU are determined to be eligible for the study and parents consent, infants will be randomized to one of 3 dose of sucrose and their pain will be assessed using a validated pain assessment measure.

ELIGIBILITY:
Inclusion Criteria:

* Infants 24 to 42 weeks gestational age (GA) at birth, admitted to the Neonatal Intensive Care Unit (NICU), and scheduled to receive a heel lance will be eligible. Parents will be approached for participation within the first 2 weeks of the infant's life. Infants will be eligible for Trial 1, the non-opioid trial, if they have not received any opioids within 24 hours prior to the heel lance. Infants will be eligible for Trial 2, the opioid trial, if they are currently receiving an opioid infusion. Furthermore, observation of the procedures will be timed to ensure that no additional sucrose doses are provided within the previous 4 hours.

Exclusion Criteria:

* Infants will be excluded if they have a contraindication for sucrose administration (e.g., unable to swallow, pharmacologically muscle relaxed, or heavily sedated) due to safety concerns and/or inability to assess pain accurately (e.g., unable to clearly view the infant's face).

Ages: 1 Day to 2 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 291 (Actual)
Dates: Start 2013-07; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
The primary outcome is pain intensity measured using the Premature Infant Pain Profile-Revised (PIPP-R). | Change from baseline 30 seconds post painful procedure
  Premature Infant Pain Profile- Revised is a validated pain measure to assess infant pain

SECONDARY OUTCOMES:
The secondary outcome is pain intensity measured using the Premature Infant Pain Profile-Revised (PIPP-R). | Change from baseline 60 seconds post painful procedure
  Premature Infant Pain Profile-Revised is a validated pain measure to assess infant pain
The secondary outcome is frequency of occurrence of adverse events. | Starting from the administration of sucrose until the end of the procedure (procedure could last on average 6 minutes) or longer if indicated.
  The potential adverse events include: heart rate >240 beats/minute or <80 beats/minute for >20 seconds, oxygen saturation <80% for > 20 seconds, no spontaneous respirations for > 20 seconds, and choking or gagging.

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie Stevens, RN, PhD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Stevens B, Yamada J, Campbell-Yeo M, Gibbins S, Harrison D, Dionne K, Taddio A, McNair C, Willan A, Ballantyne M, Widger K, Sidani S, Estabrooks C, Synnes A, Squires J, Victor C, Riahi S. The minimally effective dose of sucrose for procedural pain relief in neonates: a randomized controlled trial. BMC Pediatr. 2018 Feb 23;18(1):85. doi: 10.1186/s12887-018-1026-x. PMID 29475433